CLINICAL TRIAL: NCT04218773
Title: A Single Center, Pilot Study of Induced Hypertension for Minimizing Infarct Progression in Patients With Acute Large-vessel Occlusion Ischemic Stroke Undergoing Endovascular Therapy
Brief Title: Blood PREssure Augmentation in Large-vessel Occlusion Stroke Study
Acronym: PRESS
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: seeking additional funding
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Nils Petersen, Assistant Professor of Neurology, Yale University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2000022525
Record Dates: First submitted 2019-12-20; First posted 2020-01-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Blood Pressure
Keywords: Induced hypertension; Blood pressure augmentation; Large-vessel occlusion; Thrombectomy; Endovascular therapy
MeSH Terms: conditions — Ischemic Stroke | interventions — Phenylephrine; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Induced hypertension (Experimental): The scientists will investigate the potential consequences of increasing baseline systolic blood pressure with intravenous fluids and phenylephrine by 20% to at least 160 mmHg until blood vessel recanalization is achieved or the thrombectomy procedure is completed. The maximum allowed SBP is 220 mmHg or 180 mmHg, if intravenous TPA was administered.
  Interventions: Drug: Phenylephrine; Drug: Norepinephrine

INTERVENTIONS:
Drug: Phenylephrine — Patients will receive intravenous phenylephrine at a rate of 60 µg/min. The infusion rate will be adjusted at 30 µg/min increments (maximum 180 µg/min) at 3-minute intervals to maintain an increase in SBP to the target SBP of 160 - 220 mmHg or a 20% increase above baseline SBP values.
  Other Names: Neo-Synephrine
Drug: Norepinephrine — As an alternative to intravenous phenylephrine, intravenous norepinephrine can be used with an initial infusion rate of 3 mcg/min. The initial infusion rate of norepinephrine will be adjusted at 1 mcg/min increments at 3-minute intervals to achieve and maintain the target blood pressure. Maximum dose is 25 mcg/min. Combination therapy with both agents (phenylephrine and norepinephrine) to achieve and maintain blood pressure targets is not permitted.
  Other Names: Levophed

SUMMARY:
An open label, prospective, single center, pilot trial to assess feasibility and tolerability of short term blood pressure augmentation to minimize infarct progression in acute LVO stroke patients undergoing endovascular therapy.

DETAILED DESCRIPTION:
The trial is planned to include 40 subjects with acute LVO stroke who meet the eligibility criteria. In stage 1 of the study, the investigators will monitor beat-to-beat blood pressure and other hemodynamic parameters in 20 patients receiving standard of care therapy. For the second stage, the investigators will enroll an additional 20 patients who will receive blood pressure augmentation therapy using intravenous fluids and phenylephrine or norepinephrine infusion. The investigators will increase baseline systolic blood pressure by 20% to at least 160 mmHg until blood vessel recanalization is achieved or the thrombectomy procedure is completed. The study will assess how quickly a target blood pressure can be reached in the acute stroke setting, and furthermore the ability to successfully maintain these blood pressure targets throughout the intervention and avoid hypotension during conscious sedation or general anesthesia. The primary research hypothesis of the trial is that treatment failure defined as an inability to achieve and maintain blood pressure targets despite the use of maximum tolerable doses of vasopressors (phenylephrine or norepinephrine) occurs in less than 20% of cases. In addition, the study will evaluate the recruitment feasibility and preliminary safety of blood pressure augmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥18 years
2. Patients presenting with anterior circulation acute ischemic stroke
3. Enrollment within 24 hours of stroke onset
4. Treatment with endovascular thrombectomy
5. Arterial occlusion on CTA or MRA of the ICA, M1 or M2
6. Mismatch - Using CT or MRI with a Tmax >6 second delay perfusion volume and either CT-rCBF or DWI infarct core volume.

   1. Mismatch ratio of greater than 1.8, and
   2. Absolute mismatch volume of greater than 15 ml, and
   3. Infarct core lesion volume of less than 70 mL

Exclusion Criteria:

1. Baseline SBP>200 mm Hg
2. Intracranial hemorrhage (ICH) identified by CT or MRI
3. Inability to access the cerebral vasculature in the opinion of the neurointerventional team
4. Contraindication to imaging with MR
5. A history of a left ventricular heart failure (NYHA Class ≥ III, or EF < 50%) or angina (either unstable or CCS Grade II) involving symptoms at rest or with ordinary physical activity
6. Acute myocardial infarction in the past 6 months
7. Signs or symptoms of acute myocardial infarction, including electrocardiogram find-ings, on admission
8. Elevated serum troponin concentration on admission (>0.1 μg/L)
9. Suspicion of aortic dissection on admission
10. Participation in any investigational study in the previous 30 days
11. Treatment with Monoamine oxidase inhibitors (MAO-I) within last 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Outcome: Ability to achieve and maintain systolic blood pressure goals | Through completion of the thrombectomy procedure, an average of 2.5 hours
  Percentage of treatment success is defined as the percentage of patients able to achieve target blood pressure within 60 minutes and maintain it throughout the procedure.
Primary Safety Outcome: Number of patients with symptomatic intracranial hemorrhage | 72 hours
  Symptomatic intracerebral hemorrhage (sICH) is defined per SITS-MOST criteria as local or remote parenchymal hemorrhage type 2 on the post-treatment imaging scan, combined with a neurological deterioration of 4 points or more on the NIHSS from baseline, or from the lowest NIHSS value between baseline and 24 h, or leading to death.

SECONDARY OUTCOMES:
Total number of serious adverse events | 24 hours
  Number of treatment-related SAEs including but not limited to myocardial infarction, congestive heart failure and death during the first 24 hours from enrollment. Any SAE judged probably or definitely related to the study treatment is counted as a treatment-related SAE. The timeframe for SAE is based on the rapid onset and short half-life of phenylephrine and norepinephrine. Late SAEs are not expected to be related to treatment; however, these SAEs also are ascertained.

OTHER OUTCOMES:
Recruitment feasibility: Rate of patient identification | Though study completion, an average of one year
  Rate of patient identification will be calculated as the number of eligible patients who were identified and approached for consent by the study team divided by the number of eligible patients.
Recruitment feasibility: Rate of consent | Though study completion, an average of one year
  Patient rate of consent will be calculated as the number of eligible patients who provided consent for participation divided by the total number of eligible patients.
Recruitment feasibility: Enrollment rate | Though study completion, an average of one year
  Patient enrollment rate will be calculated as enrolled patients per month.
Recruitment feasibility: Time to enrollment | Though study completion, an average of one year
  Time to enrollment will be assessed by calculating the time from ED presentation to enrollment in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nils H Petersen, MD, MSc, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No